CLINICAL TRIAL: NCT07234604
Title: Is 3D Modeling From Non-contrast CT Accurate for Minimally Invasive Lung Segmentectomies ?
Acronym: 3D-LS
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9776
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer
Keywords: Lung cancer; Segmentectomy; 3D reconstruction; Computed tomography; Minimally invasive surgery
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical stage IA lung lesions & malignancy: Patient with clinical stage IA lung lesions ≤ 2 cm in diameter AND a suspected or proven malignancy, cf eligibility criteria
  Interventions: Diagnostic Test: Thoraco-abdomino-pelvic CT scan without and with contrast injection.

INTERVENTIONS:
Diagnostic Test: Thoraco-abdomino-pelvic CT scan without and with contrast injection. — Eligible patients undergo the usual preoperative procedure, including consultations and CT scan with and without contrast injection.

SUMMARY:
To assess the RELIABILITY in terms of accuracy of 3D-CT and 2D-CT reconstructions compared to intraoperative data regarding bronchovascular anatomy and tumor location. 3D CT reconstruction (CT scan without contrast injection) with Innersight3D® is equivalent to 2D CT (CT scan with contrast injection) for planning a minimally invasive lung segmentectomy.

Evaluate the impact of 3D reconstruction (from a CT scan without injection of contrast agent) on intraoperative and postoperative results

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥ 18 years
* Patient agreeing to participate in the study
* Patient with clinical stage IA lung lesions ≤ 2 cm in diameter AND a suspected or proven malignancy.
* Chest CT scan available without and then with contrast
* Eligible for VATS or RATS segmentectomy based on respiratory explorations

Exclusion Criteria:

* Patient refusal to participate in the study
* Allergic reactions to radiographic contrast agents
* History of ipsilateral cardiothoracic surgery
* Open segmentectomy (thoracotomy)
* Histology different from that of NSCLC
* Inability to provide the subject with informed information (difficulty understanding the subject, insufficient command of French, etc.)
* Pregnant or breastfeeding women
* Severe cognitive impairment and/or suspicion of lack of compliance or adherence, in the investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adult patient ≥ 18 years
  * with clinical stage IA lung lesions ≤ 2 cm in diameter AND a suspected or proven malignancy.
  * Chest CT scan available without and then with contrast
  * Eligible for VATS or RATS segmentectomy based on respiratory explorations
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
RELIABILITY of 3D-CT and 2D-CT reconstructions regarding bronchovascular anatomy and tumor location - composite 1 | Immediately after surgery
  Accuracy between predicted bronchovascular anatomy by 3D CT and 2D CT reconstruction compared to intraoperative observations
RELIABILITY of 3D-CT and 2D-CT reconstructions regarding bronchovascular anatomy and tumor location - composite 2 | Immediately after surgery
  Accuracy between predicted tumor location by 3D CT and 2D CT reconstruction compared to intraoperative observations

CONTACTS AND LOCATIONS:
Locations (1):
- Service Chirurgie Thoracique - CHU de Strasbourg - France, Strasbourg, Strasbourg, France